CLINICAL TRIAL: NCT03807414
Title: Development of a Web-based Multicenter Registry on the Use of oXiris Membrane for Extracorporeal Blood Purification Therapies in Critically Ill Patients
Brief Title: Development of a Web-based Multicenter Registry on the Use of oXiris Membrane for EBPTs in Critically Ill Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Careggi Hospital (Other)
Collaborators: University of Florence (Other)
Responsible Party: Principal Investigator, Gianluca Villa, Principal investigator, Careggi Hospital
Other Study IDs: CEAVC14334
Record Dates: First submitted 2019-01-08; First posted 2019-01-16 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Critical Illness; Acute Kidney Injury; Sepsis; Systemic Inflammatory Response Syndrome
Keywords: intensive care unit; regisrty; endotoxin; heparin
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury; Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Critically ill patients: In centres that obtained IRB approval for this prospective study, all critically ill adult patients (>18yrs) undergoing treatment with oXiris will be prospectively observed.
  Interventions: Device: oXiris

INTERVENTIONS:
Device: oXiris — Every center will prescribe EBPT with oXiris in accordance with local practice and local levels of expertise. No variation in treatment prescription and/or treatment solutions will derive from participation in this prospective observational study. Nonetheless, every setting parameter will be recorded in the web-based registry and analyzed a-posteriori to reveal a potential correlation with the patient outcomes.

SUMMARY:
The use of extracorporeal blood purification therapies (EBPT) is becoming increasingly widespread worldwide in everyday clinical practice, particularly in the critical care setting. Nonetheless, most of the clinical trials aimed at exploring the effect of EBPT on patients' long-term outcomes have failed to demonstrate consistent results regarding 28 day- or hospital- mortality rates. The aim of this observational prospective registry is to evaluate if there is a cluster of critically ill patients that mostly benefits from extracorporeal blood purification therapies with oXiris membrane.

DETAILED DESCRIPTION:
The use of extracorporeal blood purification therapies (EBPT) is becoming increasingly widespread worldwide in everyday clinical practice, particularly in the critical care setting. For most of these treatments, the extracorporeal removal of inflammatory mediators (via enhanced transmembrane clearance and/or selective/un-selective adsorption of bacterial toxins or inflammatory mediators) is already well established in the literature. Unselective cytokine removal is the main rationale for the use of EBPT, and it might explain the effect of these treatments on multiorgan dysfunction in critically ill patients. Indeed, an increment in hemodynamic stability and an improvement in the multiorgan dysfunction scoring system of treated patients are consistently observed in most of the studies available in the literature. Nonetheless, most of the clinical trials aimed at exploring the effect of EBPT on patients' long-term outcomes have failed to demonstrate consistent results regarding 28 day- or hospital- mortality rates.

Interestingly, the post-hoc analysis of large databases suggests that a specific subpopulation of patients, who are likely to benefit more than others from EBPT, could be identified in clinical practice. As an example, press releases from the Euphrates trial suggest that a specific range of baseline endotoxin activity assay might correlate with a positive long-term outcome in patients treated with Toraymixin cartridges. Nowadays, a personalized approach to extracorporeal therapy has been advocated as the only strategy capable of maximizing the clinical effect of EBPT and their impact on patient outcomes (i.e. precision medicine).

The identification of clinical characteristics correlated with positive outcomes during EBPT allows the implementation of specifically designed trials, focused on a well-defined cluster of patients.

The implementation of a large database encompassing the clinical/biochemical characteristics of patients undergoing EBPT is thus widely hoped for to enable the identification of a cluster of patients with specific features who most benefit from these treatments.

Although it is well known that only a clinical trial can formally assess the effect of EBPT on a specific clinical outcome, several drawbacks pose practical limitations to the implementation of a clinical trial in the critical care setting for this purpose. First, most European countries (and particularly Italy) do not allow the enrollment and randomization of non-competent patients (as critically ill patients formally are), due to ethical issues. Second, clinical trials are associated with very high costs. Third, the quality of results and conclusions deriving from post-hoc analysis of randomized clinical trials (often underpowered) may be qualitatively similar to those obtained from a very large database of patients observed during treatments performed according to the routine clinical practice.

As an example, COMPACT and COMPACT 2 trials, failed to demonstrate a significant effect of Coupled plasma-filtration adsorption (CPFA) on the outcome of critically ill septic patients, with the notable exception of specific subpopulations (e.g. those where an adequate volume of plasma was filtered and adsorbed). This conclusion was obtained through two highly-costly multicenter randomized clinical trials, prematurely halted due to ethical issues, using post-hoc analysis of a subgroup of an already limited sample size.

Nowadays, the identification of specific clusters of patients during EBPT is obtained by means of the implementation of a large web-based registry where a network of researchers can upload the clinical data of patients undergoing EBPT in line with the routine clinical practice of each single center. Taking into consideration the feasibility of the research (i.e. mainly related with the lack of critical ethical issues and the easy-to-use interface of web-platforms), these observation-based registries are inexpensive and effective tools able to identify specific clusters of patients within a very large sample size with widely heterogeneous clinical characteristics.

As an example, a web-based registry has been already implemented to describe the clinical effects of polymyxin-B based cartridges for endotoxin removal (EUPHAS 2 registry). Another one has been similarly implemented to describe the clinical effects of un-selective cytokine adsorption obtained with CytoSorb (CytoSorb registry).

Taking into consideration the fact that data on CPFA already exist and web-based registries are already available for Toraymixin and for CytoSorb, the aim of this project is to design and nationally promote a web-based registry specifically designed for oXiris membrane. In particular, an easy-to-use web-based platform will be made available for all centers that spontaneously adhere to this project.

Three main characteristics will distinguish this web-based registry of the clinical use of oXiris membrane when compared with the already available Euphas 2 and CytoSorb registries. First, it will also be available for smartphone and/or tablet applications; this characteristic will guarantee easy-to-use access and data uploading and enhanced compliance from clinical researchers. Second, it will not be confined to a simplistic registration of patients' data; it will instead also provide the clinician with clinical tools that might be helpful for patient management (e.g. automatic calculation of clinical scoring systems, ideal body weight, functions of mechanical ventilation, antibiotic adjustment according to renal function, etc.). All these tools will provide the clinician with real-time feedback; this web-based registry will provide a clear example of translational medicine and translational research, where data from clinical practice will feed a database for clinical research and, contemporaneously, the research tool will improve clinical practice, providing useful instruments for routine practice. Finally, this web-based registry will allow every center to instantaneously evaluate its results, providing a real-time basic statistic for every recorded variable (e.g. age at enrollment, main comorbidities, baseline serum creatinine, mortality rate, rate of multidrug resistant bacteria, etc.). This function may allow each center to continuously monitor outcomes and local practices, and will represent a major improvement when compared to already existing platforms in Italy, such as the Prosafe.

With this rationale, the research questions are:

* Is there a cluster of critically ill patients that mostly benefits from extracorporeal blood purification therapies (EBPT) with oXiris membrane?
* Might some baseline variables be used to identify this subpopulation of "responsive" patients? In particular, may these indicators be employed to guide indications for EBPT with oXiris, in order to personalize treatments and improve patients' long-term outcome?

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients in the ICU
* treatment with oXiris

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All critically ill patients undergoing EBPT with oXiris membrane in the enrolling centers will be prospectively observed.
  Although acute kidney injury will be mostly present among the enrolled population, it will be not strictly required as an inclusion criterion. Similarly, although sepsis will be frequently observed, the systemic inflammatory state leading to multiorgan dysfunction and supported by these extracorporeal treatments might have several different etiologies, such as ischemia-reperfusion, severe acute pancreatitis, intoxication, etc. (i.e. "sepsis-like syndromes").
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Identification of the subpopulation of critically ill patients that most benefits from EBPT with oXiris | 10 days after EBPT initiation
  This subpopulation will be described using the baseline variables associated with a positive long-term patient's outcome. In particular baseline variables statistically associated through multivariable regression analyses with the patient's survival at hospital discharge will be identified and expressed with their Odds ratios, 95%CI and p-value

SECONDARY OUTCOMES:
Description of the over-time variation of clinical variables during EBPT with oXiris. | 24 hours after EBPT initiation
  This over-time variation will be expresed, for each variable, as a percentage variation compared with the baseline value (at the EBPT initiation).

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Villa, MD, Principal Investigator — U. of Florence- Dept of Health Sciences
Locations (12):
- Italy (12):
  - Presidio Ospedaliero di Esine, Esine, Brescia
  - S. Giuseppe Hospital, Empoli, Firenze
  - IRCCS Policlinico S. Donato Milanese, San Donato Milanese, Milano
  - Ospedale Sacro Cuore di Gesù-Fatebenefratelli, Benevento
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - A.O.U. della Campania "L. Vanvitelli", Napoli
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale S. Maria della Misericordia, Perugia
  - Ospedale San Jacopo, Pistoia
  - S.Camillo Forlanini Hospital, Roma
  - Cristo Re Hospital, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cruz DN, Antonelli M, Fumagalli R, Foltran F, Brienza N, Donati A, Malcangi V, Petrini F, Volta G, Bobbio Pallavicini FM, Rottoli F, Giunta F, Ronco C. Early use of polymyxin B hemoperfusion in abdominal septic shock: the EUPHAS randomized controlled trial. JAMA. 2009 Jun 17;301(23):2445-52. doi: 10.1001/jama.2009.856. PMID 19531784
- [Background] Klein DJ, Foster D, Schorr CA, Kazempour K, Walker PM, Dellinger RP. The EUPHRATES trial (Evaluating the Use of Polymyxin B Hemoperfusion in a Randomized controlled trial of Adults Treated for Endotoxemia and Septic shock): study protocol for a randomized controlled trial. Trials. 2014 Jun 11;15:218. doi: 10.1186/1745-6215-15-218. PMID 24916483
- [Background] Livigni S, Bertolini G, Rossi C, Ferrari F, Giardino M, Pozzato M, Remuzzi G; GiViTI: Gruppo Italiano per la Valutazione degli Interventi in Terapia Intensiva (Italian Group for the Evaluation of Interventions in Intensive Care Medicine) is an independent collaboration network of Italian Intensive Care units. Efficacy of coupled plasma filtration adsorption (CPFA) in patients with septic shock: a multicenter randomised controlled clinical trial. BMJ Open. 2014 Jan 8;4(1):e003536. doi: 10.1136/bmjopen-2013-003536. PMID 24401721
- [Background] Cutuli SL, Artigas A, Fumagalli R, Monti G, Ranieri VM, Ronco C, Antonelli M; EUPHAS 2 Collaborative Group. Polymyxin-B hemoperfusion in septic patients: analysis of a multicenter registry. Ann Intensive Care. 2016 Dec;6(1):77. doi: 10.1186/s13613-016-0178-9. Epub 2016 Aug 8. PMID 27502196
- [Background] Friesecke S, Trager K, Schittek GA, Molnar Z, Bach F, Kogelmann K, Bogdanski R, Weyland A, Nierhaus A, Nestler F, Olboeter D, Tomescu D, Jacob D, Haake H, Grigoryev E, Nitsch M, Baumann A, Quintel M, Schott M, Kielstein JT, Meier-Hellmann A, Born F, Schumacher U, Singer M, Kellum J, Brunkhorst FM. International registry on the use of the CytoSorb(R) adsorber in ICU patients : Study protocol and preliminary results. Med Klin Intensivmed Notfmed. 2019 Nov;114(8):699-707. doi: 10.1007/s00063-017-0342-5. Epub 2017 Sep 4. PMID 28871441
- [Derived] Villa G, Fioccola A, Cecchi M, Scire Calabrisotto C, Pomare Montin D, De Rosa S, Scoccia G, Manno A, Tofani L, Santorsola C, Patera F, Capitanini A, Resta MV, Ferrari F, Greco M, Rossi F, Ricci Z, Ronco C, Romagnoli S; OxirisNET registry working group. Use of Oxiris membrane in real-world clinical practice in critical care patients: a multicenter observational study. J Anesth Analg Crit Care. 2025 Dec 15;5(1):91. doi: 10.1186/s44158-025-00305-3. PMID 41398301
- [Derived] Santorsola C, Corona A, Cecchi M, Nicolini NC, Zendra E, Capone A, Gatti I, Brivio M, Falsini S, Villa G. Dynamic CRRT Prescription for Complicated Critically Ill Patient: A Case Report. Case Rep Crit Care. 2024 Nov 20;2024:1837150. doi: 10.1155/2024/1837150. eCollection 2024. PMID 39611098